CLINICAL TRIAL: NCT02211534
Title: A Randomized, Sham-Controlled Pilot Study of Pulsed Electromagnetic Field Therapy in the Treatment of Persistent Post-Operative Pain Following Total Knee Arthroplasty
Brief Title: Pilot Study of PEMF Therapy in Treatment of Post-operative Pain Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBI.2014.002
Record Dates: First submitted 2014-08-01; First posted 2014-08-07 (Estimated); Results first posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Post-Operative Pain Following Total Knee Arthroplasty
Keywords: Pulsed Electromagnetic Energy Fields; Total Knee Arthroplasty; Pain Intensity
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulsed Electromagnetic Field Device (Active Comparator): Pulsed Electromagnetic Field therapy device; self-administered at home twice daily for 30 minutes.
  Interventions: Device: Pulsed Electromagnetic Field Device (Provant)
- Sham Pulsed Electromagnetic Field Device (Sham Comparator): Inactive Pulsed Electromagnetic Field Therapy device; self-administered at home twice daily for 30 minutes.
  Interventions: Device: Sham Pulsed Electromagnetic Field Device

INTERVENTIONS:
Device: Pulsed Electromagnetic Field Device (Provant) — The PEMF device delivers non-thermal, non-ionizing pulsed electromagnetic energy to the target tissue, using 27.12 megahertz pulses lasting 42 microseconds and delivered 1000 times per second. The system generates an electromagnetic field that is continuously monitored and regulated to ensure consistent dosing. The therapeutic electromagnetic field is delivered by means of an applicator pad that is placed against the treatment site. The active and sham devices will be identical in appearance and all other physical characteristics in order to maintain the masking of the treatment.
  Other Names: Provant Therapy System
  Arms: Pulsed Electromagnetic Field Device
Device: Sham Pulsed Electromagnetic Field Device — The Sham device will be identical in appearance, physical characteristics and operation to the Active device.
  Other Names: Sham Provant Therapy System
  Arms: Sham Pulsed Electromagnetic Field Device

SUMMARY:
The purpose of this study is to investigate whether pulsed electromagnetic energy field (PEMF) therapy is effective in the treatment of persistent pain following total knee arthroplasty (TKA)

DETAILED DESCRIPTION:
This is a multi-site randomized, double-blinded, parallel-group prospective pilot study of the analgesic effectiveness of twice-daily PEMF therapy in the treatment of persistent post-operative pain following Total Knee Arthroplasty (TKA). Following a run-in period of 10 days to collect their baseline pain intensity scores, activity levels and opioid consumption, eligible subjects will be randomized in a 2:1 ratio to receive therapy with an active PEMF device or an identical inactive Sham device. Subjects will self-treat twice daily for 60 days while at home. Subjects will collect electronic patient-reported outcome (ePRO) data each morning through Day 75. Subjects will be evaluated at the research center for Interim Visits at Day 21, Day 41, Day 61 and Day 75 for assessment of safety, concomitant medications, range of motion, weight, peripheral edema, and quality of life outcomes. At Day 90, Day 150, and Day 240 assessment of pain intensity, opioid consumption, safety, review of concomitant medications and interval history will be performed, with data collected via telephone contact.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater or equal to 18 years.
2. Subject has undergone a total knee replacement for the treatment of osteoarthritis, and has persistent post-operative pain in the index knee for > 3 months and < 36 months following surgery.
3. Subject has been receiving medication for persistent post-operative knee pain, including opioid or non-opioid analgesic medication that is administered on an "as needed" (prn) basis, and is on a stable analgesic dosing regimen (i.e. the same medications and dosages) for > 30 days prior to the screening visit.
4. Mean Pain Intensity (calculated as the mean of the daily average pain intensity scores) is ≥3 and < 9 as measured on Numeric Pain Rating Scale (NPRS) during the run-in phase.
5. Subject has completed a minimum of 80% (8 of 10 possible) of the pain intensity assessments during the run-in phase.
6. Subject is willing and able to wear an activity meter from the screening visit through Day 75.
7. Subject is able to access an internet browser in the home environment.
8. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.
9. Female Subjects must be post menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject has undergone simultaneous bilateral knee arthroplasty or revision arthroplasty on the index knee.
2. Subject requires revision surgery prior to Day 75.
3. Subject has undergone manipulation under anesthesia of the index knee or any local injection into the index knee within 30 days prior to the Screening Visit, or within 6 weeks prior to the Screening Visit for long acting lidocaine injection products.
4. Subject has received any investigational drug or device within 30 days prior to the Screening Visit or is enrolled in another clinical trial.
5. Subjects consuming an average of > 100 mg oral Morphine Sulfate equivalents per day during the run-in phase.
6. Subject has evidence on physical or radiological exam of joint instability or infection involving the index knee.
7. Passive range of motion demonstrates maximal flexion of the index knee < 90 degrees or maximal extension of the index knee < -10 degrees.
8. Body Mass Index (BMI) < 19 kg/m2, or > 38 kg/m2.
9. Subject has a history of any uncontrolled medical illness that in the investigator's judgment places the subject at unacceptable risk for receipt of Provant therapy.
10. Subject has an ongoing painful condition that in the opinion of the Investigator might have a confounding influence on the safety or effectiveness analysis for this study.
11. Use of systemic corticosteroids within 2 months of the Screening visit.
12. Subject anticipates the need for surgery of any type through the Day 75 visit.
13. Subjects whom, in the judgment of the Investigator, have serious psychosocial co-morbidities.
14. History of drug or alcohol abuse within one year prior to screening.
15. Subject has a history of malignancy within the past five years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area and/or localized carcinoma in situ of the cervix.
16. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
17. Existing or planned pregnancy.
18. Subject has been previously treated with study device.
19. Subject is in current litigation related to the index knee or is receiving Worker's Compensation for an injury related to the index knee.
20. Subject is unwilling or unable to follow study instructions, comply with the treatment regimen, study visits, and ePRO assessments.
21. Standard deviation around the mean of the average pain intensity scores during the run-in period is >2.0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - El Cajon, California
  - Lone Tree, Colorado
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Las Vegas, Nevada
  - New York, New York
  - Raleigh, North Carolina
  - Spartanburg, South Carolina
  - St. George, Utah
  - Danville, Virginia
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Started | 24 | 11
Completed | 11 | 6
Not Completed | 13 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device | Total
Number analyzed (Participants) | 24 | 11 | 35
Age, Continuous [Mean (Full Range); unit: Years] | 62.42 [45 to 76] | 63.82 [45 to 79] | 62.86 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 7 | 24
  Male | 7 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 21 | 10 | 31
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 10 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Pain Catastrophizing Score [Mean (Full Range); unit: units on a scale] — The Pain Catastrophizing Scale (PCS) is a validated assessment tool for the extent to which patients catastrophize their pain. The scale asks 13 questions about types of thoughts and feelings associated with pain. Responses are based upon a 5-point scale ranging from 0 to 4, where 0=not at all and 4=all the time. A total score is calculated ranging from 0 to 52. Higher scores represent a higher catastrophization of pain.
  The PCS will be administered at the research center during the Screening Visit, and scored by research personnel.
  units on a scale | 19 [0 to 45] | 17.7 [0 to 40] | 18.59 [0 to 45]
BMI [Mean (Full Range); unit: kg/m^2] | 31.3 [23.2 to 36.9] | 31.7 [28 to 38] | 31.42 [23.2 to 38]
PainDETECT Questionnaire [Mean (Full Range); unit: units on a scale] — PainDETECT Questionniare (PD-q): a self-reported assessment designed to identify the presence of a neuropathic pain component in subjects with pain. Subjects assessed current pain, strongest pain, average pain, areas of pain, course of pain and symptoms (such as burning, tingling, numbness and sensitivity). The scale ranged from 0 to 38 defined as follows: score 0-12 = neuropathic pain component unlikely; 13-18 = result is ambiguous; 19-38 = neuropathic pain component is likely.
  units on a scale | 12.8 [4 to 31] | 12.7 [1 to 26] | 12.8 [1 to 31]

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity
Description: Percent change from Baseline in Pain Intensity (PI): a validated 11-point Numeric Pain Rating Scale (NPRS) with scores (0-10) collected as patient-reported outcomes on an electronic diary (ePRO). A score of 0 represents 'No Pain' while a score of 10 represents "Worst Pain Imaginable".
Time Frame: Assessed at Day 60 as compared to Baseline
Population: Discrepancy in Numbers of Participants Analyzed is due to the number of subjects completing the Day 60 assessment. Not all subjects that were enrolled and had baseline data captured completed the Day 60 assessment. Subjects without a Day 60 assessment were left out of the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 22 | 10
Units on a scale | -30.9 (37.99) | -29.7 (30.58)

2. Secondary Outcome: Mean Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: Knee Injury and Osteoarthritis Outcome Score (KOOS): a validated knee-specific instrument that measures the short-term and long-term symptoms and function associated with knee injury. KOOS consists of 5 categories: pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life. Patients are asked to answer questions relating to these categories and respond with Never/None/Not at all, Rarely/Monthly/Mild, Sometimes/Moderate/Weekly, Often/Severe/Daily or Always/Extreme/Totally/Constantly. Each response gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The mean change in score from baseline to Day 75 is displayed below.
Time Frame: Mean change from Day 0 to Day 75
Population: Discrepancy in Numbers of Participants Analyzed is due to the number of subjects completing the Day 75 assessment. Not all subjects that were enrolled and had baseline data captured completed the Day 75 assessment. Subjects without a Day 75 assessment were left out of the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 22 | 10
units on a scale | 9.2 (19.02) | 8.9 (14.17)

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Responders: Defined as subjects with a 5-point decrease in Beck Depression Inventory (BDI) score.
  BDI is a validated self-reported assessment of current symptoms of depressive disorders, with total scores ranging from 0 to 63. The BDI scale consists of 21 groups of statements with each score/response ranging from 0 to 3. Higher scores represent greater depression. The BDI was conducted at baseline prior to study device treatments and again at Day 61.
Time Frame: Responders at Day 75 (compared to baseline)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 22 | 10
Participants | 3 | 2

4. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Responder Analysis at Day 75 (patents stating they are "Improved" to "Much Improved") using the Patient Global Impression of Change (PGIC). PGIC is a 7-point validated categorical scale of overall change in status since initiation of treatment with the study device. PGIC allows subjects to integrate into one overall evaluation the different aspects of their response to treatment, including pain reduction, improvement in functioning and side effects. Subjects select one of the following response at the end of treatment: Very Much Worse, Much Worse, Minimally Worse, No Change, Minimally Improved, Improved, or Much Improved.
Time Frame: Day 75
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 22 | 10
Participants | 5 | 2

5. Secondary Outcome: Analgesic Consumption
Description: Consumption of opioid analgesics in the preceding 24 hours will be self-reported by the subject in the ePRO diary on a daily basis during the 10-day run-in period, treatment period and through Day 75. The results below display the difference in opioid analgesic consumption from baseline to Day 56-60. Subject recorded the number of tablets consumed.
Time Frame: Day 56 to Day 60 (compared to baseline)
Population: Number of Participants Analyzed differs from numbers above due to the number of subjects reporting opioid analgesic consumption in their ePRO diary.
Measure: Mean (Standard Deviation); unit: Number of tablets taken
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 10 | 4
Number of tablets taken | -20.6 (18.04) | -22.2 (16.78)

6. Secondary Outcome: Change From Baseline in Range of Motion (ROM)
Description: The degree of passive (movement of the knee with the aid of study personnel) and active (subject moving the knee) knee flexion and extension tolerated by the subject will be recorded. ROM will be assessed in the sitting position using a goniometer.
Time Frame: Days 0 (Baseline) and Day 75
Measure: Mean (Standard Deviation); unit: degrees of motion
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 21 | 9
degrees of motion
  Change from Baseline - Passive Extension ROM-Day75 | -.5 (3.72) | .4 (3.09)
  Passive Extension ROM - Baseline | 3.2 (2.81) | 3.6 (4.13)
  Active Extension ROM - Baseline | 4.4 (3.37) | 4.2 (3.8)
  Change from Baseline - Active Extension ROM-Day75 | -.8 (3.49) | .6 (2.4)
  Change from Basline - Passivie Flexion ROM-Day 75 | 3.0 (9.19) | 4.6 (4.93)
  Passive Flexion ROM - Baseline | 110.3 (11.44) | 110.0 (16.05)
  Active Flexion ROM - Baseline | 107.7 (10.35) | 106.8 (14.85)
  Change from Baseline - Active Felexion ROM -Day 75 | 3.7 (9.19) | 5.2 (7.69)

7. Secondary Outcome: Change From Baseline in Peripheral Edema - Maximal Circumference of Calf (cm)
Description: The maximal circumference of the calf and circumference of the thigh at 10 cm and 15 cm cranial to the superior pole of the patella of the index knee will be measured using a tape measure.
Time Frame: Day 75
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 21 | 9
cm | .1 (1.46) | -.1 (0.75)

8. Secondary Outcome: Change in Pain Intensity - Average Pain Intensity
Description: Pain Intensity (PI): a validated 11-point Numeric Pain Rating Scale (NPRS) with scores (0-10) collected as patient-reported outcomes on an electronic diary (ePRO).
Time Frame: At Days 75, 90, 150 and 240, as compared to Baseline
Population: Data were not collected.
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Pulsed Electromagnetic Field Device | Sham Pulsed Electromagnetic Field Device
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/11
Other Adverse Events (participants affected / at risk) | 6/24 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Electromagnetic Field Device (N=24) | Sham Pulsed Electromagnetic Field Device (N=11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Arrhythemia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated is not permitted without the prior written consent of the sponsor. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.